CLINICAL TRIAL: NCT03211923
Title: Muscle Relaxation Properties in Myopathies With Positive Muscle Phenomena: a Study Using Transcranial Magnetic Stimulation
Brief Title: Muscle Relaxation in Myopathies With Positive Muscle Phenomena
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL57301.091.16
Record Dates: First submitted 2017-06-28; First posted 2017-07-07 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2018-09

CONDITIONS: Nemaline Myopathy Type 6; Myotonic Dystrophy Type 2; McArdle Disease
Keywords: muscle relaxation; transcranial magnetic stimulation; myopathy
MeSH Terms: conditions — Myotonic Dystrophy; Glycogen Storage Disease Type V; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Nemaline myopathy type 6 (NEM6): Patients diagnosed with nemaline myopathy type 6 (mutation in KBTBD13 gene). The aim is to measure five male and five female patients.
  Interventions: Diagnostic Test: Transcranial magnetic stimulation (TMS)
- Myotonic dystrophy type 2 (DM2): Patients diagnosed with myotonic dystrophy type 2 (pathological repeat expansion in CNBP gene). The aim is to measure five male and five female patients.
  Interventions: Diagnostic Test: Transcranial magnetic stimulation (TMS)
- McArdle disease (McA): Patients diagnosed with McArdle disease (mutation in PYGM gene). The aim is to measure five male and five female patients.
  Interventions: Diagnostic Test: Transcranial magnetic stimulation (TMS)
- Healthy controls: 14 male and 10 female healthy subjects were measured in a previous study
- Controls with positive muscle phenomena: 9 male and 8 female subjects with positive muscle phenomena but no myopathy, ruled out by normal muscle biopsy, CK level, and genetic testing. These subjects were measured in a previous study.
- Brody disease: 4 male patients diagnosed with Brody disease (ATP2A1 mutation). All Dutch patients suffering from Brody disease (n=4) were measured in a previous study

INTERVENTIONS:
Diagnostic Test: Transcranial magnetic stimulation (TMS) — Single pulse, monophasic transcranial magnetic stimulation
  Groups: McArdle disease (McA); Myotonic dystrophy type 2 (DM2); Nemaline myopathy type 6 (NEM6)

SUMMARY:
The aim of this study is to quantify muscle relaxation properties of the finger flexor muscles in patients with different myopathies. The inhibiting effects of transcranial magnetic stimulation (TMS) on the cortical motor hand area are used to induce relaxation, which in turn will be monitored with handgrip dynamometry and EMG. The investigators will evaluate if this technique can be implemented as a diagnostic tool in clinical practice.

Muscle relaxation is an often overlooked property of the muscle as compared to muscle strength or activation. Muscle relaxation is affected in different myopathies, such as myotonic dystrophy, non-dystrophic myotonias, and Brody myopathy. Therefore, a diagnostic tool to quantify muscle relaxation is of clinical and scientific importance. In this study, transcranial magnetic stimulation (TMS) is used, in combination with a dynamometer to quantify muscle relaxation properties.

Transcranial magnetic stimulation (TMS) is a non-invasive technique that is commonly used to stimulate the brain. In practice, a circular coil is held directly above the scalp, upon which a strong current pulse induces a magnetic field that stimulates the underlying superficial brain areas. This stimulation can have both activating and inhibiting effects.

When the motor cortex (i.e. the area of the brain that controls muscle contractions) is strongly stimulated with TMS during a voluntary muscle contraction, both excitatory and inhibitory effects can be observed in the muscle the targeted cortical area controls. The inhibitory effect entails a transient interruption of neural drive to the muscle. This interruption, called the "silent period", lasts for less than half a second and results in the relaxation of the muscle. Muscle activity and control quickly return to normal after the silent period.

The elegance and main advantage of TMS-induced muscle relaxation lies in the fact that it excludes all voluntary influences on the relaxation process. Furthermore, the TMS pulse causes all muscle fibres involved in the contraction just prior to the onset of the silent period to relax simultaneously. This allows us to study muscle relaxation as only a property of the muscle, i.e. without voluntary influences.

In this study, the investigators will measure muscle relaxation in several myopathies (McArdle disease, Nemaline myopathy type 6 and myotonic dystrophy type 2) and compare this to healthy controls and to controls with no myopathy but with similar complaints (myalgia, stiffness, cramps). The data from these two control groups has been gathered previously in a different study. The investigators will also compare this to patients suffering from Brody disease who were previously measured in a different study.

Muscle relaxation will be evaluated in fresh and fatigued finger flexor muscles. The main outcome of this study is the peak relaxation rate normalized to the peak force preceding relaxation.

The final outlook of this research is to evaluate whether muscle relaxation studied with TMS, can be used for different myopathies as a diagnostic tool, to monitor disease progression, and to study the effects of different interventions (e.g. medication, exercise).

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of one of the following myopathies: Nemaline myopathy type 6 (NEM6), Myotonic dystrophy type 2 (DM2), McArdle disease.

Exclusion Criteria:

* Pregnancy
* Serious head trauma or brain surgery
* Large or ferromagnetic metal parts in the head
* Implanted cardiac pacemaker or neurostimulator
* Epilepsy, convulsion or seizure
* Use of medication that can influence muscle relaxation or cortical excitability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of one of the following myopathies: Nemaline myopathy type 6 (NEM6), Myotonic dystrophy type 2 (DM2), McArdle disease.
  Patients will be selected from a local database at the Radboud University Medical Center. The goal is to include 5 men and 5 women per myopathy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Normalized peak relaxation rate | 1 hour
  Maximal rate at which the muscle relaxes after the TMS pulse, defined as the steepest point on the force curve.
  This value is normalised to the force that preceded relaxation, i.e. top of the superimposed twitch.

SECONDARY OUTCOMES:
Force decline at 150ms | 1 hour
  The force decline (percentage of peak force) at 150ms after TMS stimulation.
Relaxation times (RT) | 1 hour
  The time needed for force to decline to a certain percentage of peak force. E.g. the 75% relaxation time, is defined as the time needed for force to decline from 100% (i.e. force before relaxation onset) to 75%.
  Different relaxation times will be evaluated, e.g. 90% RT, 75% RT, and 50% RT
Maximal muscle strength | 1 hour
  The highest point on the force curve prior to TMS stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Baziel G van Engelen, MD, PhD, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No